CLINICAL TRIAL: NCT00177645
Title: Inhaled Bicarbonate Therapy in Cystic Fibrosis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: Cystic Fibrosis Foundation (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 0405245
Record Dates: First submitted 2005-09-13; First posted 2005-09-15 (Estimated); Last update posted 2023-09-07 (Actual); Status verified 2016-01

CONDITIONS: Cystic Fibrosis
Keywords: cystic fibrosis; mucus clearance
MeSH Terms: conditions — Cystic Fibrosis | interventions — Sodium Bicarbonate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- sodium bicarbonate (Experimental): inhaled sodium bicarbonate
  Interventions: Procedure: sodium bicarbonate

INTERVENTIONS:
Procedure: sodium bicarbonate — inhalation of sodium bicarbonate or sodium chloride

SUMMARY:
The purpose of this study is to see if inhaled bicarbonate will increase the ability to cough up mucus in a person with cystic fibrosis.

DETAILED DESCRIPTION:
There is evidence that people with CF may have differences in the liquid that lines the surface of their lungs from people without CF. There are two things that are known to be different. One is called bicarbonate secretion, which is the movement of a salt called bicarbonate that is normally present in the blood and lung fluid in all people. The abnormal movement of bicarbonate appears to cause a second abnormality - the liquid in the breathing tubes has more acid than the liquid in patients without CF. These differences may affect the stickiness and thickness of the mucus and limit how well the hairs that line the breathing tubes (cilia) move mucus out of the lungs.

Recent studies in a group of patients with chronic cough looked at the effects of giving an inhaled bicarbonate solution (sodium bicarbonate instead of sodium chloride) on the study subjects' ability to cough up mucus. Compared to the group given inhaled saline, the patients given inhaled bicarbonate were able to cough up approximately three times as much mucus. No clinical studies have looked at whether inhaled bicarbonate improves the ability of the lung in a person with CF to move mucus out of the lung or how this treatment affects lung function in patients with CF.

ELIGIBILITY:
Inclusion Criteria:

* age 12 or older
* Forced expiratory volume in one second (FEV1) >40% predicted
* Ability to expectorate sputum

Exclusion Criteria:

* pregnancy
* pulmonary exacerbation or initiation of inhaled or oral antibiotics, steroids, or aerosol treatments within the last four weeks
* oxygen saturation <92%, or requirement for supplemental oxygen

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2002-03; Primary Completion 2006-12 (Actual); Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
Determine the acute effects of increasing doses of inhaled bicarbonate on mucociliary clearance after a single inhalation | single dose escalation

SECONDARY OUTCOMES:
comparison of pre- and post-bicarbonate exhaled breath condensate pH values at a single inhalation | two doses in single day
Safety as determined by pre- and post-clearance assay pulmonary function tests (FEV1) at a single visit | two doses in single day

CONTACTS AND LOCATIONS:
Overall Officials: Joseph M Pilewski, MD, Principal Investigator — University of Pittsburgh
Locations (1):
- Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No